CLINICAL TRIAL: NCT07204015
Title: Body Composition in Pediatric Patients With Thalassemia Major Attending Assiut University Children's Hospital
Brief Title: Body Composition in Pediatric Patients With Thalassemia Major
Acronym: BC-THAL
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Haidy Rady Gayed Hennes Saied, Principal lnvestigator, Assiut University
Other Study IDs: Body Composition,Thalassemia
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Body Composition in Thalassemia Major

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess body composition (fat mass, lean mass, and bone mass) in pediatric patients with beta thalassemia major using appropriate tools (e.g.,Bioelectrical impedance analysis (BIA)).

To evaluate the association between body composition and clinical parameters such as transfusion frequency, nutritional status, serum ferritin levels, endocrine complications.

DETAILED DESCRIPTION:
Thalassemias are severe inherited anemias characterized by microcytic, hypochromic, and short-lived red blood cells due to defective hemoglobin synthesis(1) β-thalassemias are a heterogeneous group of hereditary hemoglobinopathies characterized by defects in the β-globin chain of hemoglobin and belong to autosomal recessive disorders(2) Three clinical and hematological conditions of increasing severity are recognized and include beta-thalassemia carrier state, thalassemia intermedia, and thalassemia major (3, 4).

Regular blood transfusion is a vital treatment in β-thalassemia major patients to prevent the consequences of anemia. Iron overloading is frequently observed in β-thalassemia major patients with transfusion therapy . Excessive iron can cause multiple organ damage (5, 6, 7, 8).

Patients with β-thalassemia major (BTM) suffer from several patterns of growth retardation including short stature, underweight, wasting, and decreased bone density(9, 10).

Impaired nutritional status has been commonly observed in patients with thalassemia major. Specific nutritional deficiencies, such as vitamin D deficiency, are also often observed due to increased losses of micronutrients or increased endogenous requirements (11).

Patients suffering from thalassemia major have impaired body composition, especially whole-body lean mass and bone mineral density(12, 13). Body composition is influenced by many parameters including age, gender, endocrine system status, nutrition, and exercise (14). All the above parameters are impaired in patients with thalassemia major in addition to hyperactivity of bone marrow, iron overload, and diminished bone mineral density (15, 16).

Patients with thalassemia tend to have increased adiposity(17, 18). These alterations in body composition are more frequently seen in thalassemic patients compared to the general population and are related to the high prevalence of sarcopenic obesity (19).

Bioelectrical impedance analysis (BIA), a technique using electrical properties to analyze body composition. Using BIA provides a more accurate and non-invasive assessment of muscle mass(20).

Body composition in pediatric patients with beta_thalassemia major has not been well studied, especially in Egypt.There is a lack of sufficient data addressing changes in muscle mass, fat distribution, and their metabolic consequences in this group of patients.

This study will provide new insights into body composition profile of thalassemic children in Assisut University Children's Hospital.The results are expected to fill an important gap in knowledge, support early detection of abnormalities, and contribute to better strategies for management and prevention of long_term complications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-18 years
* Diagnosed with beta thalassemia major
* Receiving regular transfusions
* Informed consent/assent provided.

Exclusion Criteria:

* Presence of other chronic systemic diseases
* On medications that significantly affect body composition (e.g., steroids)
* Severe physical or cognitive disability interfering with assessment

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents aged 5 to 18 years with a confirmed diagnosis of beta thalassemia major attending Assiut University Children's Hospital. Both sexes will be included.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Body composition parameters (Fat Mass, Fat Free Mass) | Assessed at baseline and every 6 months for up to 12 months.
  Body composition will be assessed using bioelectrical impedance analysis (BIA) to measure fat mass, fat-free mass in pediatric patients with beta thalassemia major.

SECONDARY OUTCOMES:
Association between transfusion frequency, nutritional status, serum ferritin, endocrine complications and body composition. | Measured at baseline and every 6 months for up to 12 months
  This outcome evaluates how transfusion burden, nutritional status, iron overload (measured by serum ferritin) and endocrine complications are related to body composition in chronically transfused patients.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuriyan R. Body composition techniques. Indian J Med Res. 2018 Nov;148(5):648-658. doi: 10.4103/ijmr.IJMR_1777_18. PMID 30666990
- [Background] Visser M, van Venrooij LM, Vulperhorst L, de Vos R, Wisselink W, van Leeuwen PA, de Mol BA. Sarcopenic obesity is associated with adverse clinical outcome after cardiac surgery. Nutr Metab Cardiovasc Dis. 2013 Jun;23(6):511-8. doi: 10.1016/j.numecd.2011.12.001. Epub 2012 Mar 6. PMID 22397879
- [Background] Wong P, Fuller PJ, Gillespie MT, Kartsogiannis V, Milat F, Bowden DK, Strauss BJ. The effect of gonadal status on body composition and bone mineral density in transfusion-dependent thalassemia. Osteoporos Int. 2014 Feb;25(2):597-604. doi: 10.1007/s00198-013-2454-y. Epub 2013 Aug 1. PMID 23903954
- [Background] Fung EB, Xu Y, Kwiatkowski JL, Vogiatzi MG, Neufeld E, Olivieri N, Vichinsky EP, Giardina PJ; Thalassemia Clinical Research Network. Relationship between chronic transfusion therapy and body composition in subjects with thalassemia. J Pediatr. 2010 Oct;157(4):641-7, 647.e1-2. doi: 10.1016/j.jpeds.2010.04.064. Epub 2010 Jun 12. PMID 20547400
- [Background] Katz S, Weinerman S. Osteoporosis and gastrointestinal disease. Gastroenterol Hepatol (N Y). 2010 Aug;6(8):506-17. PMID 20978554
- [Background] Casale M, Citarella S, Filosa A, De Michele E, Palmieri F, Ragozzino A, Amendola G, Pugliese U, Tartaglione I, Della Rocca F, Cinque P, Nobili B, Perrotta S. Endocrine function and bone disease during long-term chelation therapy with deferasirox in patients with beta-thalassemia major. Am J Hematol. 2014 Dec;89(12):1102-6. doi: 10.1002/ajh.23844. Epub 2014 Sep 26. PMID 25197009
- [Background] De Sanctis V, Soliman AT, Elsedfy H, Skordis N, Kattamis C, Angastiniotis M, Karimi M, Yassin MA, El Awwa A, Stoeva I, Raiola G, Galati MC, Bedair EM, Fiscina B, El Kholy M. Growth and endocrine disorders in thalassemia: The international network on endocrine complications in thalassemia (I-CET) position statement and guidelines. Indian J Endocrinol Metab. 2013 Jan;17(1):8-18. doi: 10.4103/2230-8210.107808. PMID 23776848
- [Background] Vlychou M, Alexiou E, Thriskos P, Fezoulidis I, Vassiou K. Body Composition in Adult Patients with Thalassemia Major. Int J Endocrinol. 2016;2016:6218437. doi: 10.1155/2016/6218437. Epub 2016 Nov 10. PMID 27956899
- [Background] Lidoriki I, Stavrou G, Schizas D, Frountzas M, Fotis L, Kapelouzou A, Kokkota S, Fyntanidou B, Kotzampassi K. Nutritional Status in a Sample of Patients With beta-Thalassemia Major. Cureus. 2022 Aug 14;14(8):e27985. doi: 10.7759/cureus.27985. eCollection 2022 Aug. PMID 36120275
- [Background] Fucharoen S, Ketvichit P, Pootrakul P, Siritanaratkul N, Piankijagum A, Wasi P. Clinical manifestation of beta-thalassemia/hemoglobin E disease. J Pediatr Hematol Oncol. 2000 Nov-Dec;22(6):552-7. doi: 10.1097/00043426-200011000-00022. PMID 11132229
- [Background] Fung EB, Xu Y, Trachtenberg F, Odame I, Kwiatkowski JL, Neufeld EJ, Thompson AA, Boudreaux J, Quinn CT, Vichinsky EP; Thalassemia Clinical Research Network. Inadequate dietary intake in patients with thalassemia. J Acad Nutr Diet. 2012 Jul;112(7):980-90. doi: 10.1016/j.jand.2012.01.017. Epub 2012 May 1. PMID 22551675
- [Background] Teawtrakul N, Jetsrisuparb A, Pongudom S, Sirijerachai C, Chansung K, Wanitpongpun C, Fucharoen S. Epidemiologic study of major complications in adolescent and adult patients with thalassemia in Northeastern Thailand: the E-SAAN study phase I. Hematology. 2018 Jan;23(1):55-60. doi: 10.1080/10245332.2017.1358845. Epub 2017 Jul 31. PMID 28759343
- [Background] Chen YG, Lin CL, Ho CL, Chen YC, Kao CH. Risk of coronary artery disease in transfusion-naive thalassemia populations: A nationwide population-based retrospective cohort study. Eur J Intern Med. 2015 May;26(4):250-4. doi: 10.1016/j.ejim.2015.02.001. Epub 2015 Feb 18. PMID 25704855
- [Background] Lobo C, Angulo IL, Aparicio LR, Drelichman GI, Zanichelli MA, Cancado R; RELATH Investigators. Retrospective epidemiological study of Latin American patients with transfusional hemosiderosis: the first Latin American epidemiological study in iron overload--the RELATH study. Hematology. 2011 Sep;16(5):265-73. doi: 10.1179/102453311X13085644680302. PMID 21902889
- [Background] Fung EB, Harmatz PR, Lee PD, Milet M, Bellevue R, Jeng MR, Kalinyak KA, Hudes M, Bhatia S, Vichinsky EP; Multi-Centre Study of Iron Overload Research Group. Increased prevalence of iron-overload associated endocrinopathy in thalassaemia versus sickle-cell disease. Br J Haematol. 2006 Nov;135(4):574-82. doi: 10.1111/j.1365-2141.2006.06332.x. Epub 2006 Oct 10. PMID 17054676
- [Background] Galanello R, Origa R. Beta-thalassemia. Orphanet J Rare Dis. 2010 May 21;5:11. doi: 10.1186/1750-1172-5-11. PMID 20492708
- [Background] Rachmilewitz EA, Giardina PJ. How I treat thalassemia. Blood. 2011 Sep 29;118(13):3479-88. doi: 10.1182/blood-2010-08-300335. Epub 2011 Aug 2. PMID 21813448
- [Background] Vichinsky EP. Changing patterns of thalassemia worldwide. Ann N Y Acad Sci. 2005;1054:18-24. doi: 10.1196/annals.1345.003. PMID 16339647